CLINICAL TRIAL: NCT06915103
Title: A Case Report of NMDAR Encephalopathy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tri Dinh, Principal Investigator, Mayo Clinic
Other Study IDs: D-25-00229R1
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Anti-NMDA Receptor Encephalitis; Mature Teratoma; Paraneoplastic Syndromes
Keywords: Magnetic Resonance; Gynecologic Surgery
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Dermoid Cyst; Paraneoplastic Syndromes | interventions — Magnetic Resonance Imaging; Salpingo-oophorectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — A pelvic MRI with and without contrast was performed for evaluation of the ovary.
Procedure: Salpingo-oophorectomy — Salpingo-oophorectomy procedure was performed on the left ovary.

SUMMARY:
This case illustrates the clinical, radiologic, and histopathologic features of Anti-NMDAR encephalitis and underscores the importance of MRI in detecting ovarian teratomas when pelvic ultrasound is inconclusive.

ELIGIBILITY:
Inclusion Criteria:

* Suspected Anti-NMDA Encephalitis

Exclusion Criteria:

* Inability to consent

Ages: 34 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patient presenting to emergency department with acute psychosis, characterized by alternating episodes of catatonia and mania, regressive speech, and inappropriate behaviors.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Anti-NMDA Encephalitis | 1 week
  Diagnosis of Anti-NMDA Encephalitis based on pelvic MRI

CONTACTS AND LOCATIONS:
Overall Officials: Tri A. Dinh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No